CLINICAL TRIAL: NCT01579136
Title: Do Home Monitors Improve Blood Pressure Control?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subjects
Sponsor: Exempla Saint Joseph Hospital (Other)
Responsible Party: Principal Investigator, Karen Weber, DO, FACP, Associate Director Outpatient Services, Internal Medicine Residency Program, Exempla Saint Joseph Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201147
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): This group will not get a home blood pressure monitor.
- Home monitors (Experimental): This group will be given a home blood pressure monitor to use.
  Interventions: Behavioral: Home blood pressure monitor

INTERVENTIONS:
Behavioral: Home blood pressure monitor — The patients using home monitors checked their blood pressure on Monday, Wed, and Friday. They took 2 measurements 5 minutes apart after sitting 5 minutes in the left arm.
  Other Names: Home monitor: Omron BP760 upper arm monitor
  Arms: Home monitors

SUMMARY:
The purpose of this study is to determine if home blood pressure monitors can help decrease blood pressure in patients with diabetes at a low income clinic.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* diabetes as defined by HgA1C over 6.5%,
* uncontrolled blood pressure (SBP > 130 and or DBP > 80)

Exclusion Criteria:

* pregnancy,
* transplanted organ,
* MI/CHF/CVA within 3 months,
* dialysis,
* arrhythmia,
* metastatic cancer,
* dementia,
* visual or hearing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
change in blood pressure over time | baseline and 3 months
  We are measuring the change in blood pressure between 2 groups: the intervention group which will be using home blood pressure monitors and the control group which will get care as usual for their blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Caritas Clinic, Exempla Saint Joseph Hospital, Denver, Colorado, United States